CLINICAL TRIAL: NCT01737580
Title: Enhancing Influenza Vaccination in Seniors With TLR (Toll Like Receptor) Agonists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H12-02574
Record Dates: First submitted 2012-11-21; First posted 2012-11-29 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Influenza Vaccination in Seniors
Keywords: influenza, human; influenza vaccines; older adults; immune response
MeSH Terms: conditions — Influenza, Human | interventions — resiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intanza+resiquimod gel (Active Comparator): Intanza 15mcg intradermal injection + resiquimod gel applied to the vaccination site immediately post vaccination.
  Interventions: Drug: resiquimod
- Intanza + placebo gel (Placebo Comparator): Intanza 15mcg intradermal injection + placebo gel applied to the vaccination site immediately post vaccination.
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: resiquimod
  Other Names: R-848
  Arms: Intanza+resiquimod gel
Drug: placebo gel
  Arms: Intanza + placebo gel

SUMMARY:
The application of the TLR7/8 (Toll Like Receptor) agonist gel (immune response helper) resiquimod will enhance the immune response to the intradermal influenza vaccine in seniors 65-75 years of age.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent provided by the subject, who can be male or female
* subjects who the investigator believes can and will comply with the requirements of the protocol (i.e. return for follow-up visits, record safety observations and able to converse with study personnel including by personal telephone
* male or female age 65-75 years at visit 1
* in generally good health (stable chronic conditions acceptable), living independently or with minimal assistance (clinical frailty score 1-5) and able to attend clinic appointments
* receipt of influenza vaccination for the 2012-2013 influenza season

Exclusion Criteria:

* receipt of any live vaccine within 4 weeks or inactivated vaccine within one week of visit 1 or planned administration of any non-study vaccines between visits 1 and 2
* systemic hypersensitivity to influenza vaccine, hen's eggs or other vaccine constituent e.g. neomycin sulphate, kanamycin, formalin
* severe reaction to any previous influenza vaccine or vaccine component
* bleeding disorder, including anticoagulant therapy or thrombocytopenia, that contraindicates IM (intramuscular) injection or blood collection (does not include daily low dose ASA (acetylsalicylic acid), Plavix, and certain other mild anticoagulants with minimal bleeding risk)
* incapacity to provide fully informed consent or be attentive to follow-up observations, resulting from cognitive impairment, abuse of alcohol, or drug addiction
* lack of telephone access, inadequate fluency in English, uncertain availability during the 4 week study participation
* immune compromise resulting from disease or immunosuppressive systemic medication use within 3 months of visit 1
* receipt of blood or blood products within 3 months of visit 1
* unstable medical conditions, as indicated by a requirement for hospitalization or a substantial medication change to stabilize said condition within 3 months.
* personal frailty, determined by Clinical Frailty score of 6-7 (moderately frail or severely frail)or failure on the TUG test (Timed Up and Go time greater than 10 seconds) or inability to walk 1/4 mile, based on self report
* history of Guillain-Barre Syndrome
* psoriasis
* recent or current febrile illness with oral temperature greater or equal to 38.0 degrees centigrade or other moderate to severe illness within the previous 48 hours (may vaccinate once condition has resolved)

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Reactogenicity of the vaccine regimens | Day 0 - Day 28
  Reactogenicity of the vaccine regimens (Intanza+resiquimod gel; Intanza+placebo gel) will be collected from Day 0 (pre vaccination) to Day 7. The change from Day 0 to Day 7 will be measured. The following information will be collected and compared 1) local pain (none, mild, moderate, severe; 2) injection site redness, swelling, induration measured in millimeters; itchiness present or not 3) bruising; 4) fever-values greater than or equal to 38.0 will be considered fever; 5) general symptoms-shivering, sweating nausea, vomiting diarrhea will be measured for presence or absence; 6) general symptoms-myalgia (muscle aches), arthralgia (joint aches), malaise (feeling unwell), tiredness/fatigue, headache and sleep disturbance will be measured as mild, moderate or severe
HAI (hemagglutination inhibition)titres | Day 28 post vaccination
  The primary immunologic outcome will be the 28 day post vaccination immune (HAI, hemagglutination immune assay titer)responses to the 3 vaccine strains present in each vaccine, assessed by the EMEA/CHMP (European Medicines Evaluation/Committee on Human Medicinal Products) Agency criteria for evaluation on immune response to influenza vaccines in persons over 60 years of age. The measurements include seroconversion rate (CHMP threshold greater than 30%), geometric mean titre (GMT) fold-increase or ratio (threshold greater than 2) and seroprotection rate (threshold greater than 60%). Whether the CHMP threshold for each measurement is met or exceeded per strain will be noted between products as descriptive information.
Granzyme B levels and Interferon gamma to interleukin 10 ratios | Day 0 and Day 28 post vaccination
  The day 0 (pre vaccination) and day 28 Granzyme B levels and Interferon gamma to interleukin 10 ratios will be measured and the change in levels from Day 0 to Day 28 will be compared in the 2 groups: 1) Intanza+resiquimod gel; 2) Intanza+placebo gel

SECONDARY OUTCOMES:
Change in Microneutralization titres | Day 0 and Day 28 post vaccination
  Microneutralization titers will be measured in serum for the 3 virus strains in the influenza vaccine and compared at Day 0 (pre vaccination) and Day 28.
baseline Granzyme B Activity | Day 0 and Day 28 post vaccination
  Differences between baseline Granzyme B activity in lysates of PBMC's (peripheral blood mononuclear cells) and Granzyme B levels,interferon gamma to interleukin-10 ratios and HAI (hemagglutination inhibition) titres will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jan P Dutz, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Vancouver General Hospital, Vancouver, British Columbia, Canada